CLINICAL TRIAL: NCT01306084
Title: Viral Infections in Healthy and Immunocompromised Hosts
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110109; 11-I-0109
Record Dates: First submitted 2011-02-26; First posted 2011-03-01 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-07

CONDITIONS: Anogenital Herpes; COVID-19; Herpes Labialis
Keywords: SARS-CoV-2; Respiratory Infections; Norovirus; Adenovirus; Coronavirus; Natural History; Viral Infection; Respiratory Viruses
MeSH Terms: conditions — COVID-19; Herpes Labialis; Respiratory Tract Infections; Adenoviridae Infections; Coronavirus Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1: NIH campus employees who have recently recovered from COVID-19
- 2: Clinical Center health care workers and ancillary staff who have close patient contact and possible exposures to SARS-CoV-2
- 3: Healthy and immunocompromised subjects who have or are suspected to have a viral infection
- 4: Healthy and immunocompromised subjects exposed to someone who has a viral infection or is suspected of having a viral infection
- 5: Healthy subjects who grew up in dengue endemic areas.
- 6: Healthy subjects with a history of viral hepatitis

SUMMARY:
Background:

- Viral infections are an important cause of illness and death in hospitalized patients as well as outpatients. New strains of viruses may appear and infect both healthy people and those with weak immune systems. A better understanding of these new virus strains (such as SARS-CoV-2, the virus that causes COVID-19) may help to control and prevent these infections. In particular, some viral infections that are less problematic in healthy persons can be life threatening in persons with weak immune systems, and viruses may be able to evolve more rapidly in persons with weak immune systems and therefore develop resistance to existing treatments. Researchers are interested in collecting samples and information from otherwise healthy persons or persons with weak immune systems to study the effects of viruses and their development.

Objectives:

- To collect samples and data from individuals who have been exposed to or have contracted viral infections.

Eligibility:

* Individuals of all ages who have been diagnosed with a viral infection are suspected to have a viral infection, or have been in close contact with someone with a suspected or actual viral infection that is of interest to investigators in the Laboratory of Infectious Diseases.
* Healthy persons and persons with weak immune systems (immunocompromised individuals) are eligible to participate.

Design:

* Participants will be pre-screened to determine if they meet the eligibility criteria for the trial.
* If eligible, evaluation may include a medical chart review, a history and physical examination, review of clinical reports from outside hospitals and laboratories, and review of tissue biopsies.
* Study procedures may include collection of blood, urine, saliva, nasal fluid sampling, throat swabs, stool, and genital swabs. For participants who have specimens collected as part of their medical care (e.g. wound swabs, spinal tap, bronchoscopy, liver biopsy etc.), researchers may use leftover specimens from the clinical laboratory for testing.
* Specimens may be collected up to 4 times per week during the first 2 weeks after enrollment, and then as many as 2 times per week for up to 2 years. Some participants may be asked to continue providing specimens if there is concern for relapse or recurrence of the infection.
* Treatment is not offered under this study.

DETAILED DESCRIPTION:
Viral infections are an important cause of morbidity and mortality in hospitalized patients as well as out-patients. New strains of viruses may appear and cause epidemics in healthy persons or immunocompromised persons. A better understanding of these new virus strains may help to control and prevent these infections. Some viral infections that would otherwise be asymptomatic or cause mild disease can be life threatening in immunocompromised persons.

Immunocompromised persons often shed high titers of virus for prolonged periods of time. In the absence of a potent immune system, viruses may evolve more rapidly in their hosts.

Therefore, analysis of sequential virus specimens from these patients can provide information on virus evolution, including how resistance to antiviral agents can develop. In addition, higher titers of virus may be associated with virus mutants that are more adapted to grow in cell culture. In this protocol we will obtain specimens containing viruses from otherwise healthy or immunocompromised patients over sequential periods of time to study their nucleic acid sequences, sensitivity to antiviral agents, cell types infected by the virus, and ability to grow in cell culture. In some cases, we will review tissue biopsies or clinical reports from outside laboratories to assist with the diagnosis of virus-associated diseases. We will also record the patient s signs and symptoms, take a short history or ask patients to fill out a questionnaire, note results of any pertinent laboratory work-up, and in some cases, obtain blood to measure immune responses, isolate antibodies or virus-specific T cells, or to look for viremia. This study will include patients with viral infections and/or receiving viral vaccines. This study should provide further understanding on how viruses evolve in their natural hosts, how they become resistant to antiviral agents, how antibody responses evolve to viruses, and might allow some currently uncultivatable viruses to be grown in cell culture.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. The protocol is open to people of all ages;

     1. Only patients greater than or equal to 2 years of age can be enrolled at the Clinical Center.
     2. Patients who are less than 2 years old may be enrolled only remotely and will not be seen at the Clinical Center.
  2. a. Persons having (or be suspected of having) a viral infection that is of interest to LID investigators.

     b. Persons that are a close contact of someone who has (or is suspected of having) a viral infection that is of interest to LID investigators or is about to receive or have recently received a viral vaccine.

     c. Persons that may have had a recent viral infection that is of interest to LID investigators that has since cleared

     d. Healthy persons who will serve as controls for (a), (b), or (c) above. These persons will be 18 years of age or older and able to provide informed consent.
  3. Adults who are unable to provide initial consent may be enrolled providing procedures per Human Research Protections Program (HRPP) Policy 403 have been followed.
  4. Only subjects that are NIH employees or contractors who work at NIH will be enrolled in the COVID19 antibody cohort study on this protocol.

EXCLUSION CRITERIA

1. Patients who are unable to safely undergo study procedures and tests.
2. Patients unwilling to have samples collected and stored for future use.
3. For the healthy controls cohort: persons who are <18 years old, decisionally impaired adults, and pregnant women

Ages: 6 Months to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy or immunocompromised subjects with viral infections, or suspected of having a viral infection, or recovering from a viral infection, or a close contact of someone who has had or is suspected to have had an acute or chronic viral infection. Subjects may either be at the Clinical Center or samples may be sent to LID directly from subjects enrolled at non-NIH sites.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-03-15 (Actual)

PRIMARY OUTCOMES:
Sample collection, analysis of immune function, or review of tissue biopsies or clinical reports from outside laboratories in designated populations with viral infections, suspected of having a viral infection, recovered from a viral infection o... | open-ended
  January 2031

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Cohen JI, Dropulic L, Wang K, Gangler K, Morgan K, Liepshutz K, Krogmann T, Ali MA, Qin J, Wang J, Vogel JS, Lei Y, Suzuki-Williams LP, Spalding C, Palmore TN, Burbelo PD. Comparison of Levels of Nasal, Salivary, and Plasma Antibody to Severe Acute Respiratory Syndrome Coronavirus 2 During Natural Infection and After Vaccination. Clin Infect Dis. 2023 Apr 17;76(8):1391-1399. doi: 10.1093/cid/ciac934. PMID 36482505
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-I-0109.html